CLINICAL TRIAL: NCT01016314
Title: A Multi-Center Prospective Randomized Study to Evaluate the Efficacy of the Aspen Spinous Process System for Use in Anterior Lumbar Interbody Fusion (ALIF)
Brief Title: Efficacy of the Aspen Spinous Process System in Anterior Lumbar Interbody Fusion (ALIF)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol amended to NCT01549366 and participants rolled into study
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASP-09-001
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspen Spinous Process System (Experimental): Subjects randomized to the Aspen study arm will have the Aspen device implanted as supplemental posterior fixation only and according to the manufacturer's recommendations.
  Interventions: Device: Aspen Spinous Process System
- Pedicle Screw Fixation (Active Comparator): Subjects randomized to the pedicle screw group will have the pedicle screws implanted according to the standard procedures and practices at that institution. The procedure may be performed according to surgeon preference, including a traditional open, minimally invasive or percutaneous approach. Only pedicle screws cleared by FDA for this indication will be used in this study.
  Interventions: Device: Pedicle Screw Fixation

INTERVENTIONS:
Device: Aspen Spinous Process System — Aspen Spinous Process System is an interspinous process fixation device
  Arms: Aspen Spinous Process System
Device: Pedicle Screw Fixation — Pedicle Screws are used for the fixation of the spine
  Arms: Pedicle Screw Fixation

SUMMARY:
This is a multi-center, prospective randomized clinical study to evaluate the clinical outcome of subjects with degenerative disc disease (DDD) treated with ALIF and supplemental posterior fixation using ASPEN Spinous Process System compared to pedicle screw instrumentation.

DETAILED DESCRIPTION:
This is a multi-center, prospective randomized clinical study to evaluate the clinical outcome of subjects with DDD who are treated with ALIF and supplemental posterior fixation using Aspen compared to pedicle screw instrumentation. The study will involve up to approximately 25 investigational sites and enroll up to 156 67 subjects. The randomization ratio of two Aspen subjects to one pedicle screw subject (2:1) will be utilized.

Subjects with lumbar DDD who are candidates for ALIF at a single level will be screened for inclusion in the study. If the subject meets all of the eligibility criteria, they will be enrolled and randomized to either the Aspen or pedicle screw group. Subjects will continue to be followed by the guidelines set forth in this clinical protocol, which include: a postoperative discharge exam; six week, three month, six month, and one year post-op visits; and, concludes with a two year post-op visit. The follow-up is counted from the day of surgery. The enrollment period is expected to be approximately 12 months and subjects will be followed for 2 years post-op for the duration of the clinical investigation. The anticipated duration of the study is approximated to be 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Scheduled for an elective single level ALIF with posterior fixation
* Diagnosis of primary symptomatic DDD confirmed with appropriate imaging studies and/or positive lumbar discography
* Oswestry Disability Index (ODI) v 2.1 score >30%
* Failed at least 6 weeks of conservative care (non-surgical)/clinical signs of neurological deterioration
* No contraindications for ASPEN spinous process system (at the discretion of the investigator)

Exclusion Criteria:

* Prior lumbar fusion surgery at any level (prior discectomy and/or laminectomy allowed)
* Spondylolisthesis grade 3 or more
* Lytic spondylolisthesis
* Incompetent or missing posterior arch at the affected level (e.g. laminectomy, pars defect)
* Currently requires laminectomy at level of surgery
* Facet joints at implant level are absent or fractured
* Post-traumatic vertebral body compromise or acute fracture at implant level
* Body mass Index (BMI) > 40
* Known allergy to titanium
* Osteoporosis: SCORE (Simple Calculated Osteoporosis Risk Estimation) will be used to screen subjects who require DEXA. Subjects with T-score < -2.5 will be excluded
* Paget's disease, osteomalacia, or any other metabolic bone disease
* Use of medications or any drug known to potentially interfere with bone/soft tissue healing (e.g. chronic systemic steroids)
* Planned use of Bone Morphogenetic Protein (BMP)
* Unlikely to comply with the follow-up evaluation schedule
* Subject has recent history (less than 3 years) of chemical substance dependency or significant psychosocial disturbance that may impact the outcome or study participation
* Participation in a clinical trial of another investigational drug or device within the past 30 days
* Systemic infection such as AIDS, HIV, and active hepatitis
* Active malignancy defined as history of invasive malignancy, except if the subject has received treatment and displayed no clinical signs and symptoms for at least five years
* Pregnant or planning to become pregnant during the length of study participation
* Involvement in active litigation related to back problems at the time of screening
* Direct involvement in the execution of this protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kee Kim, MD, Principal Investigator — University of California, Davis
Locations (5):
- United States (5):
  - Pomona Valley Hospital Medical Center, Pomona, California
  - University of California, Davis, Sacramento, California
  - Kansas University Medical Center, Kansas City, Kansas
  - New York University School of Medicine, New York, New York
  - South Texas Spine, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided